CLINICAL TRIAL: NCT03204604
Title: The Brain Ketone Body Challenge Imaging Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to obtain intervention materials
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00036958
Record Dates: First submitted 2017-04-18; First posted 2017-07-02 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Alzheimer Disease
Keywords: Memory; Dietary Treatment
MeSH Terms: conditions — Alzheimer Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Challenge A - low calorie Ensure® shake Challenge B - low calorie Ensure® shake with ketone esters
Who Masked: Participant, Care Provider, Investigator
Masking Description: Visits are listed at Challenge A or Challenge B. This serves as a double blind crossover intervention for participants and clinic staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Challenge A (Experimental): Challenge A includes Cognitive testing - (FCSRT, Story Recall, BVRT, CogState One Card Learning), and PET scan with low calorie Ensure® shake containing no ketone esters. Dietary Supplement: Challenge A - low calorie Ensure®
  Interventions: Dietary Supplement: Challenge A - low calorie Ensure®; Procedure: PET Scan; Behavioral: Cognitive Testing - FCSRT; Behavioral: Story Recall; Behavioral: BVRT; Behavioral: CogState One Card Learning
- Challenge B (Experimental): Challenge B includes Cognitive testing - (FCSRT, Story Recall, BVRT, CogState One Card Learning), and PET scan with an Ensure® shake containing ketone esters. Dietary Supplement: Challenge B - Ensure® plus ketone esters (KE)
  Interventions: Dietary Supplement: Challenge B - Ensure® plus ketone esters (KE); Procedure: PET Scan; Behavioral: Cognitive Testing - FCSRT; Behavioral: Story Recall; Behavioral: BVRT; Behavioral: CogState One Card Learning

INTERVENTIONS:
Dietary Supplement: Challenge A - low calorie Ensure® — Challenge A will include a low calorie Ensure shake for the participant to drink with no ketone esters (KE).
  Arms: Challenge A
Dietary Supplement: Challenge B - Ensure® plus ketone esters (KE) — Challenge B will include an Ensure shake for the participant to drink with deltaG ketone ester, which has generally recognized as safe (GRAS) supplement status .
  Arms: Challenge B
Procedure: PET Scan — Subject will drink the shake. Immediate recall memory testing. Subject will be placed in the scanner. Prior to PET acquisition, a low dose CT scan of the head will be obtained for attenuation correction. Patients will be injected with an intravenous bolus of up to 5-10mCi (370 MBq) (+/- 10%) of [11C]AcAc (over 2 minutes). This is the standard dose used in published clinical studies using [11C]AcAc. The PET acquisition will begin immediately after the tracer injection and last for a total of 30 minutes. 2 ml of blood will be sampled from the forearm vein at 3, 6, 8, 12, 20, and 28 minutes post [11C]AcAc tracer injection. This will be used for quantification of radiation estimates throughout the scan-period
Behavioral: Cognitive Testing - FCSRT — The Free and Cued Selective Reminding Test (FCSRT) measures verbal memory through multiple trials of a list learning task. A list of 16 items is visually presented to the participants, who then recall as many items as possible. On subsequent trials, participants are told only those items they omitted on the previous trial. The procedure continues until the participant recalls all items on two subsequent trials. After approximately 30-minute delay, participants are asked to recall as many items as possible. The number of items recalled after the delay is then summed.
Behavioral: Story Recall — Story Recall: This test is a modification of the episodic memory measure from the Wechsler Memory Scale-Revised (WMS-R). In this modified version, free recall of one short story that consists of 44 bits of information will be elicited immediately after it is read aloud to the participant and again after a thirty-minute delay. The total bits of information from the story that are recalled immediately (maximum score = 44) and after the delay interval (maximum score = 44) are recorded. Six comparable versions of this task have been validated in prior studies with older adults.
Behavioral: BVRT — Benton Visual Retention Test (BVRT): The BVRT is a multiple-choice visual recognition task. Participants view a visual pattern and are then asked to select the target from an array of four patterns, three of which are distractors. It assesses visuospatial working memory. This recognition format has the advantage assessing visual memory while eliminating the influence of visuomotor and manual dexterity difficulties.
Behavioral: CogState One Card Learning — The One Card Learning Test involves a visual learning task sensitive to early-stage cognitive impairment. It is one of several computerized assessments developed by CogState that assess executive function and working memory.

SUMMARY:
The Brain Ketone Body Challenge Imaging Study will measure how the brain uses different fuels. To do this, radioactive compounds will be used during Positron Emission Tomography (PET) imaging.

These compounds, called [11C]Acetoacetate (AcAc) and [18F] Fludeoxyglucose (FDG), are similar to the sugars and fats the brain already uses for fuel. These compounds safely allow researchers to see how the brain uses sugars and fats during PET scans.

DETAILED DESCRIPTION:
After consuming a chilled 4 ounce shake which contains various dietary fats, cognitive testing and dual-tracer Positron Emission Tomography scan will be completed. At Visit 1, each participant will be randomized to Challenge A (low calorie Ensure®) or Challenge B (Ensure® plus ketone esters). At Visit 2, each participant will undergo the remaining challenge (A or B) prior to the second imaging session. Each visit is designed to be identical to the other and only vary the dose of ketone esters. Randomization to either Challenge at Visit 1 will ensure that test/re-test learning effects are equally distributed between the challenge groups. This study consists of two visits that will take place over a two week period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Mild Cognitive Impairment (MCI)
* Stable medical condition
* Stable on medications for past 4 weeks
* Women must be post-menopausal

Exclusion Criteria:

* Diagnosis of neurodegenerative illness (except for MCI)
* History of a clinically significant stroke
* Current evidence or history in past year of focal brain lesion, head injury with loss of consciousness or meeting any Diagnostic and Statistical Manual 4 (DSM-IV) criteria for major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol or substance abuse
* Diabetes that requires current use of diabetes medications
* Current use of cholesterol/lipid lowering medications
* History of epilepsy or seizure within past year
* Contraindications for imaging (e.g. claustrophobia or high prior radiation exposure)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08-08 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Primary Outcome - Brain Ketone Utilization | 2 weeks
  The relative global uptake of [11C]AcAc during Challenge B compared to Challenge A. within each individual. How the brain uses sugars and fats for fuel and who is more likely to respond to dietary treatments.

SECONDARY OUTCOMES:
Secondary Outcome - Memory Composite Score | 2 weeks
  How brain metabolism relates to the developement of memory problems. To look at memory score changes with ketone esters supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R Hughes, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No